CLINICAL TRIAL: NCT04308473
Title: Analysis of MicroBial Metabolites After Eating Refined Food
Acronym: AMBER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wilson Tang, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19-1623
Record Dates: First submitted 2020-03-02; First posted 2020-03-16 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Dietary Habits
Keywords: Gastrointestinal Microbiome; Ultra-processed Food
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Group 1 = Ultra-Processed Food Meal + Antibiotics to suppress gut flora; Group 2 = Ultra-Processed Food Meal with No Antibiotics; Group 3 = Whole Food Meal + Antibiotics to suppress gut flora; Group 4 = Whole Food Meal with No Antibiotics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: Ultra-processed Meal + Antibiotics to supress gut flora (Experimental): Subjects in Arm 1 will take antibiotics for 3 days before the meal challenge to suppress the gut flora. The antibiotics to be used are: vancomycin, 125 mg three times daily; metronidazole, 500 mg twice daily; ciprofloxacin, 500 mg twice daily; and neomycin, 1 gram three times daily. These subjects will then consume a challenge meal of ultra-processed foods.
  Interventions: Other: Ultra-processed Food Meal
- Arm 2: Ultra-processed Meal + No Antibiotics (Experimental): Subjects in Arm 2 will not take any antibiotics prior to the meal challenge. They will consume a challenge meal of ultra-processed foods.
  Interventions: Other: Ultra-processed Food Meal
- Arm 3: Whole Food Meal + Antibiotics to supress gut flora (Experimental): Subjects in Arm 3 will take antibiotics for 3 days before the meal challenge to suppress the gut flora. The antibiotics to be used are: vancomycin, 125 mg three times daily; metronidazole, 500 mg twice daily; ciprofloxacin, 500 mg twice daily; and neomycin, 1 gram three times daily. These subjects will then consume a challenge meal of whole, unprocessed foods.
  Interventions: Other: Whole Food Meal
- Arm 4: Whole Food Meal + No Antibiotics (Experimental): Subjects in Arm 4 will not take any antibiotics prior to the meal challenge. They will consume a challenge meal of whole, unprocessed foods.
  Interventions: Other: Whole Food Meal

INTERVENTIONS:
Other: Ultra-processed Food Meal — An ultra-processed diet challenge test utilizing 1) potatoes fried in highly refined and processed vegetable oil, including corn, soybean, or canola oil, with wheat and milk derivatives; 2) a beef patty sandwich containing processed American cheese, enriched refined flour, mold inhibitor, preservatives and oxidation/reduction additives such as ascorbic acid, potassium/calcium iodate, alpha-amylase, and azodicarbonamide; and 3) a beverage composed of carbonated water, high fructose corn syrup and caramel coloring. The ultra-processed challenge meal will be obtained from a local restaurant on the day of the challenge test.
  Arms: Arm 1: Ultra-processed Meal + Antibiotics to supress gut flora; Arm 2: Ultra-processed Meal + No Antibiotics
Other: Whole Food Meal — A whole food diet challenge test utilizing 1) a side salad comprised of fresh leafy vegetables, and typical whole food toppings including fresh onion, fresh tomato, fresh carrots, and raw walnuts with a pure unrefined olive oil salad dressing; 2) a legume-based main dish including chickpeas, lentils and whole grain quinoa; 3) a fresh berry-rich smoothie beverage consisting of organic blueberries, raspberries, strawberries, bananas, and fresh orange juice. The whole food challenge meal will be made by the study team from readily available commercial foods bought from local grocery stores.
  Arms: Arm 3: Whole Food Meal + Antibiotics to supress gut flora; Arm 4: Whole Food Meal + No Antibiotics

SUMMARY:
The purpose of this study is to learn more about what happens in the human body after consuming a meal that contains ultra-processed foods like hamburgers, and if this is different to what happens after consuming a meal that contains lots of whole foods, like fresh vegetables, instead.

DETAILED DESCRIPTION:
The purpose of this study is to discover more about how the human body and the bacteria living in our intestines, known as "gut flora," react to different foods a person may consume. The investigators want to know if there are differences in compounds measured in a participant's blood and urine after eating different foods. Specifically, the investigators are interested in seeing if there are differences in these compounds after eating ultra-processed foods, like hamburgers and french fries, versus eating whole foods, like fresh fruits and vegetables. The investigators also want to know if the bacteria in our intestines may change the levels of these compounds. To this end, some subjects will be asked to take antibiotics to suppress the gut flora for three days before eating the challenge meal. Suppression of gut flora is a known effect of the antibiotics used in this study. Participants will have two study visits.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 years or above.
* Able to provide informed consent and comply with study protocol
* Able to remain on a stable aspirin regimen (either on or off aspirin or aspirin products) for 1 week prior to starting study until the end of the study period.

Exclusion Criteria:

* Significant chronic illness or end-organ dysfunction, including known history of uncompensated heart failure, renal failure, pulmonary disease, hematologic diseases.
* Active infection or received antibiotics within 6 months of study enrollment.
* Use of over-the-counter probiotic within past month.
* Chronic gastrointestinal disorders.
* Intolerance to probiotic therapy.
* Allergy to vancomycin, ciprofloxacin, neomycin, metronidazole, or lactose.
* Allergy to any of the food components of the challenge meals.
* Having undergone bariatric procedures or surgeries such as gastric banding or bypass.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Serial changes in plasma and urine metabolites and biomarkers | Pre-meal (baseline) & post-meal at 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, and 6 hours
  Serial changes in plasma and urine metabolites and biomarkers
Serial changes in plasma and urine TMAO | Pre-meal (baseline) & post-meal at 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, and 6 hours
  Serial changes in plasma and urine TMAO (trimethylamine N-oxide)

CONTACTS AND LOCATIONS:
Overall Officials: W. H. Wilson Tang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang WH, Wang Z, Levison BS, Koeth RA, Britt EB, Fu X, Wu Y, Hazen SL. Intestinal microbial metabolism of phosphatidylcholine and cardiovascular risk. N Engl J Med. 2013 Apr 25;368(17):1575-84. doi: 10.1056/NEJMoa1109400. PMID 23614584
- [Background] Wang Z, Klipfell E, Bennett BJ, Koeth R, Levison BS, Dugar B, Feldstein AE, Britt EB, Fu X, Chung YM, Wu Y, Schauer P, Smith JD, Allayee H, Tang WH, DiDonato JA, Lusis AJ, Hazen SL. Gut flora metabolism of phosphatidylcholine promotes cardiovascular disease. Nature. 2011 Apr 7;472(7341):57-63. doi: 10.1038/nature09922. PMID 21475195
- [Background] Schugar RC, Shih DM, Warrier M, Helsley RN, Burrows A, Ferguson D, Brown AL, Gromovsky AD, Heine M, Chatterjee A, Li L, Li XS, Wang Z, Willard B, Meng Y, Kim H, Che N, Pan C, Lee RG, Crooke RM, Graham MJ, Morton RE, Langefeld CD, Das SK, Rudel LL, Zein N, McCullough AJ, Dasarathy S, Tang WHW, Erokwu BO, Flask CA, Laakso M, Civelek M, Naga Prasad SV, Heeren J, Lusis AJ, Hazen SL, Brown JM. The TMAO-Producing Enzyme Flavin-Containing Monooxygenase 3 Regulates Obesity and the Beiging of White Adipose Tissue. Cell Rep. 2017 Jun 20;19(12):2451-2461. doi: 10.1016/j.celrep.2017.05.077. PMID 28636934
- [Background] Koh A, De Vadder F, Kovatcheva-Datchary P, Backhed F. From Dietary Fiber to Host Physiology: Short-Chain Fatty Acids as Key Bacterial Metabolites. Cell. 2016 Jun 2;165(6):1332-1345. doi: 10.1016/j.cell.2016.05.041. PMID 27259147
- [Background] Srour B, Fezeu LK, Kesse-Guyot E, Alles B, Mejean C, Andrianasolo RM, Chazelas E, Deschasaux M, Hercberg S, Galan P, Monteiro CA, Julia C, Touvier M. Ultra-processed food intake and risk of cardiovascular disease: prospective cohort study (NutriNet-Sante). BMJ. 2019 May 29;365:l1451. doi: 10.1136/bmj.l1451. PMID 31142457
- [Background] Hall KD, Ayuketah A, Brychta R, Cai H, Cassimatis T, Chen KY, Chung ST, Costa E, Courville A, Darcey V, Fletcher LA, Forde CG, Gharib AM, Guo J, Howard R, Joseph PV, McGehee S, Ouwerkerk R, Raisinger K, Rozga I, Stagliano M, Walter M, Walter PJ, Yang S, Zhou M. Ultra-Processed Diets Cause Excess Calorie Intake and Weight Gain: An Inpatient Randomized Controlled Trial of Ad Libitum Food Intake. Cell Metab. 2019 Jul 2;30(1):67-77.e3. doi: 10.1016/j.cmet.2019.05.008. Epub 2019 May 16. PMID 31105044
- [Background] Tang ZZ, Chen G, Hong Q, Huang S, Smith HM, Shah RD, Scholz M, Ferguson JF. Multi-Omic Analysis of the Microbiome and Metabolome in Healthy Subjects Reveals Microbiome-Dependent Relationships Between Diet and Metabolites. Front Genet. 2019 May 17;10:454. doi: 10.3389/fgene.2019.00454. eCollection 2019. PMID 31164901